CLINICAL TRIAL: NCT05521646
Title: Promoting Equitable Reproductive Health: Implementing Best Practice Postpartum Contraceptive Services Through a Quality Improvement Initiative
Brief Title: Implementing Best Practice Postpartum Contraceptive Services Through a Quality Improvement Initiative
Acronym: IMPROVE-it
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Karolinska Institutet (Other)
Collaborators: The Swedish Research Council (Other Government); Forte (Industry)
Responsible Party: Principal Investigator, Elin Larsson, Associate professor, PhD, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: Dnr 2021-05962-01
Record Dates: First submitted 2022-08-25; First posted 2022-08-30 (Actual); Last update posted 2022-10-10 (Actual); Status verified 2022-10

CONDITIONS: Contraception; Immigrant; Post Partum

STUDY DESIGN:
Intervention Model Description: cluster randomized controlled trial
Who Masked: Participant
Masking Description: The participants do not know if they go to an intervention or control clinic
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): QiC implemented
  Interventions: Other: Quality Improvement Collaborative
- Control (No Intervention)

INTERVENTIONS:
Other: Quality Improvement Collaborative — Explore if a Quality Improvement Collaborative can increase the proportion of immigrant women who choose an effective postpartum contraceptive method
  Arms: Intervention

SUMMARY:
Immigrant women in Europe has reported lower use of effective contraception, higher risks of multiple births, and unintended pregnancies compared to native-born women. There is no evidence about this from a Swedish context nor about postpartum contraception.

The purpose of this project is to promote equity in sexual and reproductive health (SRH) in Sweden by improving the quality of postpartum contraceptive counselling for and with immigrant women.

The Swedish Pregnancy Registry (SPR) will be used to determine if there are any differences in birth spacing and associated complications when comparing immigrant and Swedish-born women. Registration of contraceptive methods in the SPR will be introduced. The IMPROVE-it project will increase the understanding of challenges to contraceptive services postpartum, and how to overcome these.

DETAILED DESCRIPTION:
This cRCT will be conducted at MHCs in the regions of Jönköping, Västra Götaland and Stockholm. The unit of randomization will be the clinics. The Swedish pregnancy Register (SPR) will be used to collect data on the women's choice of postpartum contraceptive method, and the proportion of women choosing an effective method will be compared between control and intervention clinics. A survey will be completed for both groups at the postpartum visit at MHCs within 16 weeks postpartum to evaluate the choice of contraceptive method and the counselling received, as well as six and 12 months after the visit to determine ongoing contraceptive use and satisfaction with the method. Furthermore, the follow up at six and 12 months will identify any unintended or planned pregnancy, abortion, or miscarriage that has happened since the postpartum visit.

Inclusion criteria: Women coming for postpartum visit within 16 weeks post birth (live birth). Exclusion criteria: Women below 18 years or having had a still birth. The intervention clinics will register women's choice of contraception during the postpartum MHC visit and participate in Quality Improvement Collaboratives (QIC) for 12 months. The control clinics will provide routine care, register women's choice of contraception in the SPR. Recruitment: Both type of clinics will register women's choice of contraception in the SPR at the postpartum visit within 16 weeks after giving birth and ask women for consent to participate in the study, i.e. respond to a self-administered questionnaire during the visit and be contacted for follow-up. Main outcome: Proportion of women who chose an effective contraceptive method, i.e. LARC or SARC, among immigrant and Swedish-born women, as registered in the SPR at the postpartum visit within 16 weeks after giving birth.

Secondary outcomes:

At enrolment:

1. Women's satisfaction with the contraceptive counselling

   At six and 12 months after the postpartum visit:
2. Use of contraception (and type)
3. Satisfaction with the contraceptive method
4. Experiences of unintended pregnancy, abortion, miscarriages since the postpartum visit
5. Experiences of planned pregnancy since the postpartum visit

The Intervention: A QIC Initiative will be designed based on insights from the pilot study. Within the QIC, the MHCs will test evidence-based changes for contraceptive services during action periods and evaluate these during four learning seminars. Examples of evidence-based changes include using a visual aid to show contraceptive effectiveness translated to the most common languages or a person-centered counselling method based on approaches in MI and RPL. Four learning seminars will be carried out; inbetween them, there will be action periods when the midwives will test the changes made to contraceptive services in their MHC practice. Content of the learning seminars: Quality improvement methods-training; Updates on evidence-based contraceptive counselling; Feedback of data from the SPR on women's choice of contraception; Planning and evaluating tests of evidence-based changes at the MHC; Codeveloping contraceptive services in collaboration between midwives, researchers, and representatives from the target population. Part of the QIC is to continuously give data feedback to the clinics involved on women's choice of contraception. Data collection: The SPR will be used to collect and retrieve data for the primary outcome and background characteristics; a questionnaire will be used to collect data on the secondary outcome 1-2. At six and 12 months, a follow up questionnaire will be used to collect the secondary outcomes 2-5. This will be administered by SMS, email or mail. Three reminders will be sent.

Sample size and statistical power: The pilot study saw a 17% increase in the proportion of immigrant women choosing SARC/LARC. From this increase, we anticipate that at least the same share of the intervention group will be choosing SARC/LARC. Because of the cluster design, an intraclass correlation (ICC) factor affects and increases the sample size needed. The sample size was calculated to show a difference in proportions of participants choosing SARC/LARC in a two-group comparison between intervention and control groups. An assumed ICC of 0.05 was used, equivalent to the ICC observed in a similar study. To show the anticipated 15% difference in SARC/LARC choice with a 90% power at an α=0.05 (i.e. the probability of falsely rejecting a true null hypothesis), we need to include 14-15 clinics in each of the control and intervention groups, each contributing with an average of 100 participants. We will include a total of 29 clinics to allow for dropouts of clinics. The sample size calculations were performed by using the package clusterPower version 0.6.111 in R version 3.6.1. No power calculation was performed for secondary outcomes. Analysis: The analysis population will consist of all women in the cRCT. The primary analysis for the main outcome will be undertaken on an 'intention-to-treat' basis, i.e. all women with a recorded outcome will be included in the analysis and analyzed according to the group to which they were allocated, i.e. the proportion of women choosing SARC/LARC between our two randomized groups. We will further estimate the effect of the QIC using logistic regression analysis. Odds Ratios with 95% confidence intervals will be generated. A multivariate analysis will be performed to control for age, sociodemographic characteristics, and reproductive history.

ELIGIBILITY:
Inclusion Criteria:

* Women coming for postpartum visit within 16 weeks post birth (live birth)

Exclusion Criteria:

* Women who do not anticipate becoming sexually active with a male partner within six months.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 4000 (Estimated)
Dates: Start 2022-09-05 (Actual); Primary Completion 2023-09 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Proportion of women who chose an effective contraceptive method, i.e. LARC or SARC, among immigrant and Swedish-born women. | 12 months
  Data collection as registered in the Swedish pregnancy register at the postpartum visit within 16 weeks after giving birth.

SECONDARY OUTCOMES:
Womens satisfaction with the contraceptive counselling provided at the postpartum visit | 12 months
  Data collection through a questionnaire (electronic, paper or by telephone together with an interpreter if needed) filled in by the participants (electronic or paper) or by a researcher (telephone).
Participants´ use of contraception (and type) at six and 12 months follow-up | 18-24 months
  A follow-up questionnaire will be used. Data collection through a questionnaire (electronic, paper or by telephone together with an interpreter if needed) filled in by the participants (electronic or paper) or by a researcher (telephone). The follow-up questionnaire will be administered by SMS, email or mail.
Participants´ satisfaction with the contraceptive method at six and 12 months follow-up | 18-24 months
  A follow-up questionnaire will be used. Data collection through a questionnaire (electronic, paper or by telephone together with an interpreter if needed) filled in by the participants (electronic or paper) or by a researcher (telephone). The follow-up questionnaire will be administered by SMS, email or mail.
Participants´ experiences of unintended pregnancy, abortion, miscarriages since the postpartum visit, at six and 12 months follow-up | 18-24 months
  A follow-up questionnaire will be used. Data collection through a questionnaire (electronic, paper or by telephone together with an interpreter if needed) filled in by the participants (electronic or paper) or by a researcher (telephone). The follow-up questionnaire will be administered by SMS, email or mail.
Participants´ experiences of planned pregnancy since the postpartum visit, at six and 12 months follow-up | 18-24 months
  A follow-up questionnaire will be used. Data collection through a questionnaire (electronic, paper or by telephone together with an interpreter if needed) filled in by the participants (electronic or paper) or by a researcher (telephone). The follow-up questionnaire will be administered by SMS, email or mail.

CONTACTS AND LOCATIONS:
Locations (1):
- Karolinska Inst., Stockholm, Sweden

REFERENCES:
- [Derived] Kilander H, Sorcher R, Berglundh S, Petersson K, Wangborg A, Danielsson KG, Iwarsson KE, Branden G, Thor J, Larsson EC. IMplementing best practice post-partum contraceptive services through a quality imPROVEment initiative for and with immigrant women in Sweden (IMPROVE it): a protocol for a cluster randomised control trial with a process evaluation. BMC Public Health. 2023 May 3;23(1):806. doi: 10.1186/s12889-023-15776-8. PMID 37138268